CLINICAL TRIAL: NCT04778982
Title: A Phase II Study to Evaluate Efficacy, Safety and Tolerability of KN026 in Combination With Palbociclib and Fulvestrant in Patients With Locally Advanced HER2-positive Breast Cancer
Brief Title: Study of KN026 in Combination With Palbociclib and Fulvestrant in Patients With Advanced Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Difficulty in completing enrollment within the planned time
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: KN026-205
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: HER2-positive Metastatic Breast Cancer
Keywords: KN026; palbociclib; HER2-positive MBC
MeSH Terms: interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA and single cell sequencing analysis may be performed using plasma samples collected from subjects at baseline and upon disease progression.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- dose-escalation Phase: KN026 20 mg/kg + palbociclib125 mg/day+Fulvestrant 500 mg (Patients with HR+/HER2-positive MBC )
- parallel-group expansion Phase: KN026 20 mg/kg + palbociclib +Fulvestrant 500 mg(Patients with HR+/HER2-positive MBC )
  Interventions: Drug: KN026 combined with Palbociclib and Fulvestrant

INTERVENTIONS:
Drug: KN026 combined with Palbociclib and Fulvestrant — HR+/HER2-positive MBC will be treated by KN026 20 mg/kg+Palbociclib+fulvestrant 500 mg
  Other Names: combination
  Groups: parallel-group expansion Phase

SUMMARY:
This is an open-label, multicenter, dose-escalation and parallel-group expansion Phase II clinical trial to evaluate the efficacy, safety and tolerability of KN026 in combination with palbociclib and fulvestrant in women or male with HER2-positive metastatic breast cancer .The subjects will receive 20 mg/kg IV Q2W+ palbociclib 100/125 mg/day orally+/-Fulvestrant 500 mg IM until progressive disease, unacceptable toxicity or death.

DETAILED DESCRIPTION:
KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, leading to a dual HER2 signal blockade.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >= 18 years;
* Histologically or cytologically confirmed, metastatic or locally advanced unresectable HER2-positive;
* Adequate organ function assessed within 7 days prior to first trial treatment
* ECOG score 0 or 1;
* Left ventricular ejection fraction (LVEF) ≥ 50% at baseline;
* Life expectancy >3 months

Exclusion Criteria:

* Untreated active CNS metastasis or leptomeningeal metastasis;
* Uncontrolled tumor-related pain;
* Has received other anti-tumor treatment or an investigational drug within 28 days or within 5 times of half-life (whichever is shorter, and no less than 2 weeks) prior to the first trial treatment;
* Major surgery for any reason within 28 days;
* Curative radiation within 3 months of the first dose of trial treatment;
* History of uncontrolled intercurrent illness;
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosing locally advanced unresectable or metastatic HER2-positive
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 24 weeks
  The proportion of patients experiencing dose limiting toxicities
Objective response rate (ORR) | through study completion, an average of 1 year
  ORR as assessed by the investigator according to RECIST 1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | through study completion, an average of 1 year
  clinical response time (DOR) as determined by investigators based on RECIST 1.1 criteria
Progression free survival (PFS) rates | 6 months and 12 months
  Progression free survival (PFS) rates
Overall survival (OS) | 6 months and 12 months
  Overall survival (OS) rates
Clinical benefit rate (CBR) | CBR calculated as the proportion of subjects with best overall response of CR, PR, or SD ≥24 weeks
  Clinical benefit rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China